CLINICAL TRIAL: NCT03381846
Title: Treatment of Dermatofibrosarcoma Protuberans in Patients 10 Years and Younger
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Randall K. Roenigk, Professor of Dermatology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-010617
Record Dates: First submitted 2017-11-09; First posted 2017-12-22 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Dermatofibrosarcoma Protuberans
MeSH Terms: conditions — Dermatofibrosarcoma | interventions — Mohs Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MOHS treatment arm (Experimental): Patients who have their dermatofibrosarcoma protuberans excised with MOHS surgery.
  Interventions: Procedure: MOHS micrographic surgery; Procedure: Wide local excision

INTERVENTIONS:
Procedure: MOHS micrographic surgery — Mohs surgery is a precise surgical technique used to treat skin cancer. Thin layers of cancer-containing skin are progressively removed and examined microscopically until only cancer-free tissue remains.
Procedure: Wide local excision — A surgical technique in which the skin cancer is excised along with 2-3 cm of clinically normal appearing surrounding tissue.

SUMMARY:
The purpose of this proposed study is to assess effectiveness of MOHS micrographic surgery as a form of treatment for dermatofibrosarcoma protuberans in patients who are 10 years of age or younger through review of the patients at Mayo Clinic treated from 1988-2017, and to explore the challenges that providers face which may prevent them performing this potentially superior treatment. This study will provide a comparison of outcomes and recurrence rates in pediatric patients treated by MOHS versus traditional excision.

ELIGIBILITY:
Must be 10 years of age or younger. Must have biopsy proven dermatofibrosarcoma protuberans.

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Patient developing recurrence of a biopsy-proven dermatofibrosarcoma protuberans at one year. | Recurrence will be assessed at 1 year.
  Developing an additional dermatofibrosarcoma protuberans at any location, but particularly noting local recurrence (defined as being within or contiguous to the field of the previous excision.

SECONDARY OUTCOMES:
All cause mortality | All cause mortality will be assessed at 1 year, and then annually thereafter for up to 10 years. All patients will have at least one year of follow up.
  Death secondary to any cause
Mortality related to dermatofibrosarcoma protuberans | Mortality related to dermatofibrosarcoma protuberans will be assessed at 1 year, and then annually thereafter for up to 10 years. All patients will have at least one year of follow up.
  Death which is directly related to the dermatofibrosarcoma or complications related to it as judged by clinical investigators
Morbidity secondary to surgical procedure | Morbidity secondary to surgical procedure will be assessed at 1 year, and then annually thereafter for up to 10 years. All patients will have at least one year of follow up.
  Will be measured by the area of tissue removed and any functional or physical impairment which resulted from the surgical procedure such as limited range of motion, resulting reported pain, or any reported complications.
Patient developing recurrence of a biopsy-proven dermatofibrosarcoma protuberans at two years. | Recurrence will be assessed at 2 years. (Not all patients will have a full two years of follow up)
  Developing an additional dermatofibrosarcoma protuberans at any location, but particularly noting local recurrence (defined as being within or contiguous to the field of the previous excision.
Patient developing recurrence of a biopsy-proven dermatofibrosarcoma protuberans at five years. | Recurrence will be assessed at 5 years. (Not all patients will have a full five years of follow up)
  Developing an additional dermatofibrosarcoma protuberans at any location, but particularly noting local recurrence (defined as being within or contiguous to the field of the previous excision.

CONTACTS AND LOCATIONS:
Overall Officials: Randall K Roenigk, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials